CLINICAL TRIAL: NCT03165539
Title: The Effect of Intraoperative Cerebral Oxygen Desaturation on Post-Operative Delirium in Thoracic Surgical Patients: A Pilot Study
Brief Title: Cerebral Oxygen Desaturation and Post-Operative Delirium in Thoracic Surgical Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Other Study IDs: B2013:084
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Delirium; Thoracic Surgery
Keywords: Postoperative; One-lung ventilation; Cerebral oximetry; Cerebral desaturation
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Thoracic surgery patient: Pre-operatively, patients will have baseline cognitive assessment done using the Mini-mental status test and MOCA test. Intra-operatively patients' baseline cerebral saturation (%) will be measured, and continuously monitored throughout the procedure. Post-operatively, patients will be assessed for delirium using the CAM score.
  Interventions: Device: Cerebral oxygen saturation monitoring

INTERVENTIONS:
Device: Cerebral oxygen saturation monitoring — Intraoperatively, patients will have baseline cerebral oxygen saturation monitoring while breathing room air. Cerebral oxygen saturation monitoring will continue throughout the entire operation including the time on one-lung ventilation.

SUMMARY:
This study will assess the incidence and risk factors for post-operative delirium in patients undergoing thoracotomy. Specifically, the study will assess if there is any relationship between an intra-operative decrease in brain oxygen levels which can occur during one-lung ventilation, and the occurrence of delirium in the post-operative period.

DETAILED DESCRIPTION:
This will be a prospective, observational study on 200 patients. Consenting thoracic surgical patients presenting for open thoracotomy or VATS will be assessed pre-operatively for baseline cognitive status and clinically relevant risk factors for delirium. Intra-operatively, patients will undergo cerebral oxygenation monitoring using near infra-red spectroscopy cerebral oximetry. Postoperatively, patients will be assessed twice daily for the presence or absence of delirium using the Confusion Assessment Methodology (CAM) scoring system during their hospital stay.

A clinically relevant desaturation will be defined as a 25% decrease from the patient's baseline saturation, which will be determined while the patient is breathing room air pre-operatively. The severity and duration of any desaturation will be recorded and subsequently analyzed for correlation with post-operative delirium. Bivariate associations between the risk of delirium and predictor variables will be sought. If appropriate, logistic regression models will be constructed with the outcome of delirium.

Significance: Previous studies at our centre have resulted in over 35% of thoracic surgical patients developing significant, intra-operative cerebral desaturation. We propose to study a convenience sample of 200 consecutive patients. Depending on the relative risk of developing delirium with a significant cerebral desaturation, this study may be adequately powered to determine the associated risk of delirium. This study will provide background information in planning further interventional trials to prevent desaturation and possibly reduce the incidence of delirium, as well as aid in the planning of larger multi-center trials to more accurately assess the risk of intra-operative decreases in cerebral oxygenation and the role this event contributes to the occurrence of delirium.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a thoracic surgical procedure with one-lung ventilation.

Exclusion Criteria:

* Inability to communicate in English
* Lack of informed consent

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thoracic surgery patients at a major healthcare centre with a requirement for one-lung ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Post-operative Delirium vs Cerebral Desaturation | 5 days
  Incidence of delirium will be assessed post-operatively up to POD 5 as measured by positive Confusion Assessment Method (CAM) scores and correlated with clinically relevant cerebral desaturation (greater than a 25% decrease from baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jacobsohn, MD, Study Chair — University of Manitoba
Locations (1):
- Department of Anesthesia, University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vasilevskis EE, Han JH, Hughes CG, Ely EW. Epidemiology and risk factors for delirium across hospital settings. Best Pract Res Clin Anaesthesiol. 2012 Sep;26(3):277-87. doi: 10.1016/j.bpa.2012.07.003. PMID 23040281
- [Background] Berry MF, Onaitis MW, Tong BC, Harpole DH, D'Amico TA. A model for morbidity after lung resection in octogenarians. Eur J Cardiothorac Surg. 2011 Jun;39(6):989-94. doi: 10.1016/j.ejcts.2010.09.038. Epub 2011 Jan 26. PMID 21276728
- [Background] Schoen J, Meyerrose J, Paarmann H, Heringlake M, Hueppe M, Berger KU. Preoperative regional cerebral oxygen saturation is a predictor of postoperative delirium in on-pump cardiac surgery patients: a prospective observational trial. Crit Care. 2011;15(5):R218. doi: 10.1186/cc10454. Epub 2011 Sep 19. PMID 21929765
- [Background] Suehiro K, Okutai R. Duration of cerebral desaturation time during single-lung ventilation correlates with mini mental state examination score. J Anesth. 2011 Jun;25(3):345-9. doi: 10.1007/s00540-011-1136-1. Epub 2011 Apr 12. PMID 21484501
- [Background] Tang L, Kazan R, Taddei R, Zaouter C, Cyr S, Hemmerling TM. Reduced cerebral oxygen saturation during thoracic surgery predicts early postoperative cognitive dysfunction. Br J Anaesth. 2012 Apr;108(4):623-9. doi: 10.1093/bja/aer501. Epub 2012 Feb 5. PMID 22311364